CLINICAL TRIAL: NCT03021811
Title: EUREKA Italy - The Evaluation of Real-life Use of KLOX BioPhotonic System in Chronic Wounds Management: a Reproducibility Study
Brief Title: EUREKA Italy - Evaluation of Real-life Use of KLOX BioPhotonic System in Chronic Wounds Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KLOX Technologies Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ORS-K1002-P001
Record Dates: First submitted 2017-01-11; First posted 2017-01-16 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Venous Leg Ulcer; Diabetic Foot Ulcer; Pressure Ulcer
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LumiHeal (Other): Treatment of chronic wounds with KLOX LumiHeal BioPhotonic System
  Interventions: Device: KLOX LumiHeal BioPhotonic System

INTERVENTIONS:
Device: KLOX LumiHeal BioPhotonic System — Real-life use of KLOX LumiHeal BioPhotonic System in combination with standard of care.
  Other Names: LumiHeal

SUMMARY:
Multi-center, prospective, interventional, uncontrolled open-label study evaluating the real-life use of KLOX LumiHeal BioPhotonic System in chronic wounds management (venous leg ulcers, diabetic foot ulcers, pressure ulcers).

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated written informed consent form;
* Adult patient (at least 18 years old) having received a diagnosis of venous leg ulcer, diabetic foot ulcer or pressure ulcer by the Investigator;
* The treating physician (investigator) believes the KLOX LumiHeal BioPhotonic System would be an appropriate option;
* Both male and female patients must be willing to adhere to a medically-accepted birth control method during the course of the study;
* Willingness to comply with study requirements (visits, treatments, etc.).

Exclusion Criteria:

* Female pregnant patient (by medical history or as ascertained by a pregnancy test);
* Breast-feeding female patient;
* Patients taking drugs/products (e.g., methotrexate, chemotherapy agents) or with conditions (e.g., porphyria) known to induce severe photosensitivity reactions;
* Patients with known skin hypersensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Adverse events, Serious Adverse Events and Device Incidents | Up to 34 weeks
  Number of patients with adverse events, serious adverse events and device incidents.
Rate of complete wound closure | Up to 34 weeks

SECONDARY OUTCOMES:
Wound area reduction over time | Up to 34 weeks
Time to complete wound closure | Up to 34 weeks
Incidence of wound breakdown, following wound closure | Up to 34 weeks
Ease of use by healthcare professionals (questionnaire) | Up to 34 weeks
  To collect feedback on the ease of use of the KLOX LumiHeal BioPhotonic System in the management of chronic wounds, from health care professional users.
Impact of treatment on Health-related Quality of Life (CWIS questionnaire) | Up to 34 weeks
  To collect quality of life data in patients treated with the KLOX LumiHeal BioPhotonic System.